CLINICAL TRIAL: NCT07054333
Title: Objektiv Mätning av Smärtreglering Hos Personer Som Erhållit Internetförmedlad Exponeringsbaserad Kognitiv Beteendeterapi
Brief Title: Objective Measurement of Pain Regulation in Individuals Who Have Received Internet-delivered Exposure-based Cognitive Behavior Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Hedman-Lagerlöf, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-03044-01
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Within-group experimental study with participants acting as their own control.
  Participants are assessed regarding aspects of pain regulation at 10 weeks before treatment start, at treatment start (<3 days week before treatment start), at post-treatment (within 1 week of treatment completion). If we see any significant effects on any of the outcomes another assessment is made at 12 months post-treatment completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral: Internet-delivered exposure-based cognitive behavior therapy (Experimental): Internet-delivered exposure-based cognitive behavior therapy (Exp-CBT) 10-week self-help treatment delivered via a secure online platform, with regular therapist support.
  Interventions: Behavioral: Internet-delivered exposure-based cognitive behavior therapy

INTERVENTIONS:
Behavioral: Internet-delivered exposure-based cognitive behavior therapy — The primary treatment component is exposure to stimuli (situations and activities) that give rise to pain, distress, and unwanted emotional responses. The treatment proceeds in accordance with functional analysis. Exercises are tailored for the patient so that, for example, individuals whose main coping strategy is to be overly active (i.e., persistence behavior) are encouraged to sit down and observe pain and other aversive bodily sensations as they arise. The protocol also includes regular exercises where the participant is encouraged to observe and name physical sensations without acting on them.
  Other Names: Exp-CBT

SUMMARY:
Fibromyalgia: a common problem that requires treatment Fibromyalgia (FM) is a highly prevalent pain syndrome characterized by generalized pain and fatigue, often leading to extensive somatic and psychological distress. The condition is associated with significant suffering and low functional capacity, and also entails high societal costs, as those affected have high levels of healthcare consumption, sick leave, and unemployment. The cause of FM is still unclear and there is no effective treatment. The most evaluated treatment is traditional cognitive behavioral therapy (CBT), which, however, appears to have only minor effects on FM.

Exposure-based treatment promising Internet-based exposure-based CBT (Exp-CBT) has previously been evaluated for fibromyalgia in two randomized controlled studies. In the first study, participants (N=140) were randomised to 10 weeks of Exp-CBT or a waiting list. The results showed that iExp had a strong effect on central FM symptoms, pain, fatigue, function and pain-related anxiety. The study also showed that iExp, compared to no treatment, is cost-effective, and that reduced FM-related avoidance behaviors drove the treatment effect. In the second study, participants (N=274) were randomized to Exp-CBT or internet-based traditional CBT (T-CBT). The results showed no significant difference between the groups after treatment. Both groups showed a marked improvement, with an average of 60% (Exp-CBT) and 59% (T-CBT) achieving a reliable change in their symptoms. People with fibromyalgia who receive exposure-based CBT thus appear to experience, on average, a reduction in symptoms and increased function. To date, studies investigating exposure-based treatment for chronic pain have used self-assessment scales to measure the effect of treatment, which is reasonable since pain is a subjective experience. However, one limitation of this is that the investigators therefore have no objective data on whether the aforementioned treatment can also lead to changes in various aspects of pain regulation, i.e., that the brain changes the way it interprets and processes pain.

Objective measurement of pain regulation The present study is a longitudinal within-group study, in which the investigators intend to objectively measure various aspects of pain regulation in participants with fibromyalgia (N=45) before and after they have received internet-based exposure-based CBT. Participants undergo pain testing 10 weeks before (T0), at the start of treatment (T1), and at the end of treatment (T2), in order to measure the effect of treatment on participants' pain thresholds, pain tolerance, descending pain inhibitory function, and pain upregulation.

Significant potential benefits for patients, healthcare, and society In this study, the investigators want to investigate whether the investigators can objectively see if different aspects of pain regulation are affected in participants who receive the aforementioned treatment. The study is a so-called mechanistic study, i.e., a study to understand more about how our treatment achieves its effect. Such a study makes it possible to be more precise and likely to make the treatment even more effective. The study would also contribute important knowledge to better understand the pain mechanisms in fibromyalgia, a condition with high prevalence and considered very difficult to treat.

DETAILED DESCRIPTION:
Design The study is a longitudinal within-group study where participants who have received internet-delivered exposure therapy for 10 weeks are examined regarding pain regulation at 3 time points: 10 weeks before treatment start (T0), directly (within 3 days) before treatment start (T1), and directly (within 1 week) after treatment (T2). Measurements regarding subjective pain, other fibromyalgia symptoms, and function are taken weekly using electronic questionnaires from T0 to T2. Disability, fatigue, avoidance behaviors, depression, and anxiety are measured at T0, T1, and T2.

Recruitment Interested individuals are requested to register via the study's web portal where the participant receives a detailed description of the study and patient information/consent. During screening, the participant answers questions about FM symptoms, medical history, and symptoms of depression and anxiety. The Fibromyalgia Survey Questionnaire is also self-administered to evaluate diagnostic criteria and establish a diagnosis. Inclusion assessment (for inclusion and exclusion criteria, see 8.3 and 8.4) is conducted by a licensed psychologist or alternatively a psychology student under the supervision of a licensed psychologist with good knowledge in psychiatric assessment and FM. An important purpose of the assessment interview is to ensure that the potential research participants understand the study's design, as well as to ensure that participants with ongoing depression do not exhibit active suicidality by having the psychologist ask questions based on the self-assessment forms that the patients have filled out previously. Individuals who meet all criteria for participation, provide informed consent and complete the baseline assessment (T-10) are can be included in the study and scheduled for visits for pain regulation assessment and treatment (see Intervention below). The primary analysis population consists of all participants who completed the pre-measurement. Participants who withdraw their consent before the baseline assessment are not included in the analysis and are reported in the CONSORT flow as 'withdrew before baseline'.

Investigation of pain regulation

The participants will make three visits to the Karolinska Institute where different aspects of pain regulation are examined. If a significant within-group effect can be observed from pre- to post-treatment on any of the outcome measures 1-5 below, a forth assessment of pain regulation will be conducted at 12 months post treatment completion. The visits are approximately 30 min long and the examination is led by a research assistant who has been trained in the measurement procedure by Associate Professor Maria Lalouni and Professor Karin Jensen, both of whom have good knowledge in experimental pain measurement and extensive experience with the patient group. Research participants who are on pain relief medication and sleep medicine as needed are asked to refrain from using these medications 48 hours before the visits. During the visits, the following aspects of pain regulation are examined:

1. Pain threshold.
2. Pain tolerance.
3. Temporal summation (TS). Measures pain facilitation.
4. Conditioned pain modulation (CPM). Measures central, descending pain modulation according to the principle "pain inhibits pain." All above tests are conducted using two computer-controlled pressure cuffs, placed on the left and right calves (Nocitech, Denmark).
5. Lingering effect. Measures remaining pain (verbal report) 15 seconds after the tonic pain stimulation in the CPM test above has stopped.

Intervention The treatment lasts 10 weeks and is delivered through a secure web platform, where participants access self-help texts and illustrations. The texts provide the participant with the same knowledge as in conventional face-to-face treatment, and the treatment is based on the same strategies and exercises. Each module includes specific tasks that the participant must complete in order to progress in the treatment. Throughout the treatment, the participant has regular contact with a psychologist or a psychology student under supervision, who guides the participant through the treatment via text messages. The treatment manual is the same as that tested against waitlist control and traditional CBT in previous RCTs. The primary component is exposure to various situations, stimuli, and activities that the participant avoids in order to prevent pain and discomfort, combined with exercises in observing and describing bodily sensations without trying to change them. The purpose of the exercises is to increase the ability to remain in bodily discomfort and thereby facilitate the work with exposure.

Data analysis To evaluate the treatment's effect on self-report scales, data is analyzed using mixed effects regression models according to intent-to-treat. The investigators will use logistic regression to calculate the proportion of participants who achieve a clinically significant improvement (≥14% reduction on the primary outcome measure in symptom levels.

Differences in pain threshold and pain tolerance before and after treatment are measured using the Wilcoxon signed-rank test. Differences in CPM and temporal summation before and after treatment are analyzed using mixed effects regression models. Any potential association between changes in pain threshold, pain tolerance, CPM, and temporal summation on one hand and subjectively rated symptoms and adherence on the other hand will be analyzed through correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosed with fibromyalgia (indicated by a diagnosis from a physician and confirmed by the Fibromyalgia Survey Questionnaire during the assessment interview)
* Access to the internet
* Willing to refrain from other psychological treatment during the study,
* Registered with Swedish personal ID number and residing in Sweden or Finland
* If taking antidepressant or antiepileptic medication, this must be stable for 4 weeks prior to baseline measurement,
* Willing to come to Karolinska Institutet and participate in pain tests on 3-4 occasions, and
* Gives informed consent

Exclusion Criteria:

* Treatment-requiring depressive- or anxiety disorder, eating disorder or stress-related ill health, indicated by a score of ≥35 on the Montgomery-Åsberg Depression Rating Scale-Self-Rated (MADRS-S) and confirmed in a clinical assessment interview as severe depression; ongoing diagnosis of PTSD or exhaustion syndrome, unstable or unmedicated bipolar syndrome, severe obsessive-compulsive disorder or eating disorder
* Active suicidality, indicated by ≥4 on item 9 of the MADRS-S and confirmed in a clinical assessment interview
* Psychotic illness
* Late pregnancy (≥29 weeks at treatment start)
* Other somatic conditions requiring immediate treatment and/or assessed as the participant's primary problem, including other dominant pain problems and chronic fatigue syndrome (ME/CFS)
* Ongoing alcohol or substance abuse
* Opioid use
* Insufficient knowledge of Swedish or computer use to benefit from text-based treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Conditioned pain modulation | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks).
  The degree to which pain in one area of the body is reduced when a different painful stimulus is applied elsewhere. Measured by quantitative sensory testing; a test battery with various psychophysical pain tests combined with a visual analog scale. The test is performed using two computer-controlled pressure cuffs, placed on the left and right calves, for controlled induction of pain using pressure.
Pain tolerance | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks).
  Measured by quantitative sensory testing; a test battery with various psychophysical pain tests combined with a visual analog scale. The test is performed using two computer-controlled pressure cuffs, placed on the left and right calves, for controlled induction of pain using pressure.
Pain threshold | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks).
  Measured by quantitative sensory testing; a test battery with various psychophysical pain tests combined with a visual analog scale. The test is performed using two computer-controlled pressure cuffs, placed on the left and right calves, for controlled induction of pain using pressure.
Temporal summation | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks).
  The subjective pain response at repetitive pain stimulation. Measured by quantitative sensory testing; a test battery with various psychophysical pain tests combined with a visual analog scale. The test is performed using two computer-controlled pressure cuffs, placed on the left and right calves, for controlled induction of pain using pressure.

SECONDARY OUTCOMES:
Fibromyalgia severity | Screening, 10 weeks before treatment start, pre-treatment, weekly up to 10 weeks.
  The Revised Fibromyalgia Impact Questionnaire, FIQR. Self-rated, range 0-100. Higher score indicate higher FM severity.
Fatigue | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks)
  Fatigue Severity Scale, FSS. Range 9-63, higher score indicate worse outcome
Pain-related avoidance behavior | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks)
  Psychological inflexibility in pain - avoidance subscale, PIPS-avoid. Range 7-56, higher score indicate worse outcome.
Pain severity | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks)
  Severity subscale of Brief Pain Inventory-Short form (BPI-SF). Range 0-10 where higher score indicates worse outcome.
Disability | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks).
  World Health Organization disability assessment schedule 2.0, 12-item version (WHODAS 2.0). Range 0-100 where a higher score indicates worse outcome
Anxiety | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks)
  State-Trait Anxiety Inventory-State, STAI-S. Range 20-80 where higher score indicates worse outcome.
Depression | 10 weeks before treatment start, pre-treatment, post-treatment
  Beck Depression Inventory-2, BDI-2. Range 0-63 where higher score indicates worse outcome.
Lingering effect | 10 weeks before treatment start, pre-treatment, post-treatment (10 weeks)
  Verbally reported residual pain after tonic pressure pain stimulation on the non-dominant leg has been discontinued. Measured 15 s after Conditioned Pain Modulation test has been performed.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Nobels väg 9, Neuro, Stockholm, Stockholm County
  - Karolinska Institutet, Solna

IPD SHARING:
Plan to Share IPD: No
The data used in this study will not be publicly available. Reasonable requests may be directed to the principal investigator and will be considered on a case-by-case basis, in accordance with the local policies of the sponsor and the relevant Swedish and European Union data protection and privacy legislation.